CLINICAL TRIAL: NCT02077439
Title: Trial: Interactive Intention-Driven Upper-Limb Training Robotic System
Brief Title: Interactive Intention-Driven Upper-Limb Training Robotic System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Prof., The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITT/004/12GP
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Stroke
Keywords: Stroke; Hand; Upper Extremity; Robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hand Robotic Training (Experimental): Hand Robotic Training
  Interventions: Device: Hand Robotic Training
- Hand and Arm Robotic Training (Experimental): Hand and Arm Robotic Training
  Interventions: Device: Hand and Arm Robotic Training
- Conventional therapy (Active Comparator): Conventional therapy
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: Hand Robotic Training — Training for 20 sessions for one hour, 3-5 times per week.
  Arms: Hand Robotic Training
Device: Hand and Arm Robotic Training — Training for 20 sessions for one hour, 3-5 times per week.
  Arms: Hand and Arm Robotic Training
Other: Conventional therapy — Training for 20 sessions for one hour, 3-5 times per week.
  Arms: Conventional therapy

SUMMARY:
The goal of this study is to determine robotic hand system is more effective than conventional physical and occupational therapy at promoting functional recovery of the affected arm in subjects after stroke.

DETAILED DESCRIPTION:
This study will investigate the recovery in hand and upper limb functions when the physical training is assisted by an exoskeleton robotic hand system.

Subjects with a pure unilateral motor paresis after a stroke (ischemic or hemorrhagic). All subjects should have sufficient cognition to follow simple instructions as well as understand the content and purpose of the experiment, and also should be able to sit up for 1 hour.

During the training, you will be asked to do the hand open and hand grasp by Electromyography-driven robotic control strategy.

There will be evaluations on the upper limb motor functions before and after the 20-session of training and follow up session by clinical assessments on functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a pure unilateral motor paresis after a stroke (ischemic or hemorrhagic). All subjects should have sufficient cognition to follow simple instructions as well as understand the content and purpose of the experiment, and also should be able to sit up for 1 hour.

Exclusion Criteria:

* Excessive spasticity of the affected arm
* Participation in any therapeutic treatment ("outside therapy") performed with the paralyzed arm during the planned study - including baseline and follow up.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Change from baseline Fugl-Meyer Assessment at the end of intervention, at three months and at six months
  Evaluate the change from baseline assessment at the end of intervention and monitor the continuous change at three months and six months.
  Baseline assessment will be conducted at within one week prior to intervention. Participants will be followed for the duration of hospital stay, an expected average of 5 weeks for the 20-session intervention. The assessment at the end of intervention will be conducted within one week after the intervention. The other two assessments will be conducted at three months and six months after the last session of the intervention.
Action Research Arm Test | Change from baseline Action Research Arm Test at the end of intervention, at three months and at six months
  Evaluate the change from baseline test at the end of intervention and monitor the continuous change at three months and six months.
  Baseline test will be conducted at within one week prior to intervention. Participants will be followed for the duration of hospital stay, an expected average of 5 weeks for the 20-session intervention. The assessment at the end of intervention will be conducted within one week after the intervention. The other two assessments will be conducted at three months and six months after the last session of the intervention.

SECONDARY OUTCOMES:
Wolf Motor Function Test | Change from baseline Wolf Motor Function Test at the end of intervention, at three months and at six months
  Evaluate the change from baseline test at the end of intervention and monitor the continuous change at three months and six months.
  Baseline test will be conducted at within one week prior to intervention. Participants will be followed for the duration of hospital stay, an expected average of 5 weeks for the 20-session intervention. The assessment at the end of intervention will be conducted within one week after the intervention. The other two assessments will be conducted at three months and six months after the last session of the intervention.
modified Ashworth Scale | Change from baseline modified Ashworth Scale at the end of intervention, at three months and at six months
  Evaluate the change from baseline test at the end of intervention and monitor the continuous change at three months and six months.
  Baseline test will be conducted at within one week prior to intervention. Participants will be followed for the duration of hospital stay, an expected average of 5 weeks for the 20-session intervention. The assessment at the end of intervention will be conducted within one week after the intervention. The other two assessments will be conducted at three months and six months after the last session of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond KY Tong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

REFERENCES:
- See also: The Hong Kong Polytechnic University — http://www.polyu.edu.hk